CLINICAL TRIAL: NCT02271893
Title: Dextromethorphan in Chemotherapy-induced Peripheral Neuropathy Management
Acronym: CHEMODEX
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Dr Gisèle PICKERING (Unknown); Dr Dominique JOLY / Dr Christine VILLATTE (Unknown); Dr Noémie DELAGE / Dr Fabienne MARCAILLOU / Dr Pascale PICARD (Unknown); Pr Claude DUBRAY (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0214; 2014-000971-19 (EudraCT Number)
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: Chemotherapy-induced peripheral neuropathy
MeSH Terms: interventions — Dextromethorphan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Dextromethorphan (Experimental): The aim of this study is to assess if dextromethorphan administered during 4 weeks induces a decrease of pain intensity in breast cancer patients suffering from chemotherapy-induced peripheral neuropathy compared to placebo group.
  Interventions: Drug: Dextromethorphan
- placebo (Placebo Comparator): The aim of this study is to assess if dextromethorphan administered during 4 weeks induces a decrease of pain intensity in breast cancer patients suffering from chemotherapy-induced peripheral neuropathy compared to placebo group.
  Interventions: Drug: Dextromethorphan

INTERVENTIONS:
Drug: Dextromethorphan — The aim of this study is to assess if dextromethorphan administered during 4 weeks induces a decrease of pain intensity in breast cancer patients suffering from chemotherapy-induced peripheral neuropathy compared to placebo group.

SUMMARY:
The aim of this study is to assess if dextromethorphan administered during 4 weeks induces a decrease of pain intensity in breast cancer patients suffering from chemotherapy-induced peripheral neuropathy compared to placebo group.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, parallel-group clinical trial comparing dextromethorphan and placebo for the treatment of chemotherapy-induced peripheral neuropathy, assessed with a (0-10) numerical scale. Cognition, anxiety, depression, sleep and quality of life are also assessed.

The influence of CYP2D6, CYP3A4 and MDR1 polymorphism on the dextromethorphan analgesic efficacy will be measured.

ELIGIBILITY:
Inclusion Criteria:

* - Age ≥ 18 years
* Breast cancer patients suffering from chemotherapy-induced peripheral neuropathy for at least 3 months after the end of their last cancer chemotherapy
* Numerical rating scale ≥ 4
* Patient in stable clinical situation on the next month (no surgery, radiotherapy, hormone therapy, chemotherapy or other treatment scheduled in the month following the enrollment)
* Patients affiliated to the French Social Security
* Patients with free and informed consent has been obtained

Exclusion Criteria:

* - Hypersensitivity to the active substance or to any of the excipients
* Hypertension
* History of stroke
* Severe heart failure
* Severe hepatic impairment
* Shortness of breath
* Congenital galactosemia, glucose-galactose malabsorption, lactase deficiency
* Association with linezolid
* Pre-existence or history of peripheral neuropathy due to a cause different from neurotoxic chemotherapy
* Diabetes (type I and II)
* Medical and surgical history incompatible with the study
* Patient receiving treatment with amantadine, ketamine, memantine, L-Dopa, dopaminergic agonists, anticholinergics, barbiturates, neuroleptics, Monoamine oxidase inhibitor, dantrolene or baclofen, phenytoin, cimetidine, ranitidine, procainamide, quinidine, quinine, amiodarone, fluoxetine, paroxetine, propafenone, thioridazine, ritonavir, nicotine, hydrochlorothiazide, warfarin
* Present or past psychotropic substances and alcohol dependence
* Childbearing age, no use of effective contraceptive method, pregnancy or lactation
* Patient exclusion period, or the total allowable compensation exceeded
* Patients undergoing a measure of legal protection (guardianship, supervision ...)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-11-25 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
Measure of average pain intensity by a numerical rating scale | 7 days before the visit at 1 month

SECONDARY OUTCOMES:
Pain assessment by DN4 | at 1 month
total neuropathy score clinical version (TNSc) | at 1 month
St Antoine questionnaire (QDSA) | at 1 month
Evaluation of analgesic consumption | at 1 month
Cognitive assessment by Trail Making Test A and B | at 1 month
Cognitive assessment by Digit Symbol Substitution Test | at 1 month
Cognitive assessment by FACT-COG test | at 1 month
Cognitive assessment by Purdue Pegboard Test | at 1 month
Quality of life assessment by EORTC QLQ-C30 | at 1 month
Quality of life assessment by Pittsburg Sleep Quality Index (PSQI) | at 1 month
Quality of life assessment by Patient Global Impression of Change (PGIC) | at 1 month
Anxiety and Depression assessment by HAD scale | at 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Lise LACLAUTRE, Clermont-Ferrand, France

REFERENCES:
- [Derived] Martin E, Morel V, Joly D, Villatte C, Delage N, Dubray C, Pereira B, Pickering G. Rationale and design of a randomized double-blind clinical trial in breast cancer: dextromethorphan in chemotherapy-induced peripheral neuropathy. Contemp Clin Trials. 2015 Mar;41:146-51. doi: 10.1016/j.cct.2015.01.012. Epub 2015 Jan 28. PMID 25636304